CLINICAL TRIAL: NCT00769353
Title: Understanding and Treating Neuropsychiatric Symptoms of Pediatric Physical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Eva Szigethy, Associate Professor of Psychiatry, Pediatrics, and Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DP2OD001210-01 (NIH)
Record Dates: First submitted 2008-03-24; First posted 2008-10-09 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease; Depression
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy-PASCET (Experimental): Primary and Secondary Coping Enhancement Training (PASCET)
  Interventions: Behavioral: Primary and Secondary Coping Enhancement Training
- Supportive Non-Directive Therapy (SNDT) (Active Comparator): Supportive Non-Directive Therapy (SNDT)
  Interventions: Behavioral: Supportive Non-directive Therapy

INTERVENTIONS:
Behavioral: Primary and Secondary Coping Enhancement Training — A cognitive behavioral therapy designed to help individuals cope with physical illness.
  Arms: Cognitive Behavioral Therapy-PASCET
Behavioral: Supportive Non-directive Therapy — A non-structured therapy designed to provide a supportive atmosphere in which individuals may discuss concerns and process events in their lives
  Arms: Supportive Non-Directive Therapy (SNDT)

SUMMARY:
This research will examine the impact of brain activity, cognitive processing immune functioning, and gastrointestinal functioning on depressive symptoms and response to a psychotherapeutic intervention in youths with Inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
Depression is costly, worsens morbidity and mortality, and has detrimental effects on disease course in physically ill populations. This research takes a novel multi-dimensional approach to assess the neurobiological basis of depression in chronic pediatric physical illness using inflammatory bowel disease (IBD) as a model. It also evaluates the efficacy of a modified cognitive behavioral therapy (CBT) on emotional well-being, physical health, economic costs, and neurobiological outcomes. These results will provide key building blocks for a paradigm shift within medicine by integrating behavioral health into the comprehensive medical care of physical illnesses.

Little is known about how the brain and body interact to increase depressive vulnerability, particularly in youth. Adult studies identify disruptions in limbic and prefrontal brain activity in the pathophysiology of depression. Cytokines secondary to inflammation and exogenous treatment with steroids can cause mood and cognitive changes in these same brain regions. It is important to understand the neuropsychiatric effects of IBD and its treatment on underlying brain structures during adolescence, a critical developmental period for brain maturation underlying emotional regulation and cognitive processing. More importantly, neuronal plasticity during adolescence may still allow reversibility of disease-related brain effects through teaching coping strategies for life-long illness management that could change developmental trajectories and reduce vulnerability in adulthood.

Using translational neuroscience approaches, this research will examine: 1) brain regions that underlie emotional and cognitive processing in youth with active IBD and depression using brain functional magnetic resonance imaging compared to youth with IBD and no depression, and normal controls; 2) the inter-relationship between depressive symptoms in IBD and brain, immune, and gastrointestinal functioning; and 3) efficacy of a combined CBT-physical illness narrative intervention targeting emotional and cognitive processing compared to supportive non-directive therapy in the depressed IBD cohort with longitudinal tracking of emotional, physical health, economic, and neurobiological outcomes.

ELIGIBILITY:
Inclusion criteria for youths with IBD for Step 1 of Screening Process:

* Age 12 to 17 inclusive
* English-speaking
* Capable of completing CDI
* Meeting diagnostic criteria for IBD
* Absence of mental retardation by history
* Having at least one appointment at the GI clinic.

Criteria for Classification of IBD:

1. Presence of appropriate history: abdominal pain, chronic diarrhea, bloody diarrhea (with or without extraintestinal symptoms) or, less commonly, a) primary extraintestinal symptoms, b) growth retardation, c) perirectal abscess, or d) acute abdomen.
2. Evidence of colitis, ileitis or granulomatous esophagitis, gastritis or duodenitis by biopsy and/or small bowel strictures or fistulas by X-ray or multiple small intestinal ulcerations by capsule endoscopy.

Eligibility Criteria For youths with IBD for Intervention Phase of the Comparison Study

Inclusion Criteria:

1. CDI or CDI-P > 10 at Step 1
2. Childhood Depression Rating Scale-revised (CDRS-R) > 34 at Step 2
3. Presence of at least one biological parent. Exclusion Criteria

1. History or current episode of bipolar disorder, eating disorder, or psychotic disorder by Diagnostic and Statistical Manual (DSM)-IV criteria. 2. Recent suicide attempt (within 1 month of study entry) or depression severity requiring acute psychiatric hospitalization within 3 months of study entry. 3. Antidepressant medications within one month of assessment. 4. Substance abuse by history within 1 month of study entry. 5. Current treatment with CBT or failure of previous CBT trial for depression judged adequate by at least 12 treatment sessions over a period of less than 1 year conducted by an appropriately trained mental health provider using a manual. If currently receiving other psychotherapy modalities, willingness to suspend treatment for 12-week acute treatment phase of study.

Physically Healthy Comparison Children

Inclusion Criteria:

* Age 12 to 17 inclusive
* English-speaking
* Capable of completing CDI
* Absence of mental retardation by history

Exclusion Criteria:

* self-report of a cold, flu or other infection within the past two weeks
* self-reported use of any antibiotics within the past 2 weeks
* score of 6 or more on the blood draw screening questionnaire

Screening process for youths with IBD: Participants will be recruited from the clinic through a 2-step screening of all consecutive pediatric patients seen in the IBD clinic or while medically hospitalized for an IBD flare-up at Children's Hospital of Pittsburgh, who have confirmed IBD and who meet the other eligibility criteria as determined by medical staff in IBD clinic (Tables 5 and 6). The medical diagnosis of IBD will be determined by a GI physician using criteria below and will be confirmed in the medical record. Step 1: administration of the CDI and CDI-P during the medical visit. Those subjects whose CDI and/or CDI-P score of > 10 will be invited by phone to participate in Step 2: a face to face interview. Step 2 assessment will be conducted within one week of Step 1 so that both CDI score and IBD severity ratings are still valid from the Step 1 screen.

All subjects meeting eligibility criteria for Step 2 will be invited to participate in the completion of neuropsychiatric questionnaires, blood draw, pupil measurements, and brain functional magnetic resonance imaging.

All subjects meeting eligibility criteria after Step 2 will be invited to participate in the treatment phase of the study.

Normal controls (N=15) will be recruited from the Department of Pediatrics during outpatient clinical office visits.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2008-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Neurological Measures | Baseline
  Compare neurological measures (via brain scan, pupil dilation and laboratory blood values) in depressed individuals with IBD, non-depressed individuals with IBD and healthy controls.

SECONDARY OUTCOMES:
Change in baseline CDI score to three months | month 0, month 3
  Change in Childhood Depression Inventory (CDI) score from month 0 assessment to three month assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Szigethy, MD, Ph.D., Principal Investigator — University of Pittsburgh Medical Center, Children's Hospital of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391